CLINICAL TRIAL: NCT01967511
Title: Defining the Basis of Fibromuscular Dysplasia: The Define-FMD Study
Brief Title: Defining the Basis of Fibromuscular Dysplasia (FMD)
Acronym: DEFINE
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jason Kovacic, Professor, Cardiology, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 13-1118
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Fibromuscular Dysplasia; Spontaneous Coronary Artery Dissection; Cervical Artery Dissection
Keywords: Cross-sectional study; Fibromuscular dysplasia; Fibroblast; Spontaneous Coronary Artery Dissection; Cervical Artery Dissection
MeSH Terms: conditions — Fibromuscular Dysplasia; Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fibroblasts and other cell lines generated under this protocol and all blood-derived specimens (plasma, serum, DNA) will be kept indefinitely in a secure clinical database or bio-repository (as appropriate).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- FMD subjects: patients who fulfill standard diagnostic criteria for FMD
- SCAD subjects: patients who fulfill standard diagnostic criteria for SCAD
- CvAD subjects: patients who fulfill standard diagnostic criteria for CvAD
- Healthy control subjects

SUMMARY:
The purpose of this study has evolved and expanded since its inception. Originally the intent was to establish the functional, molecular and genetic profile of fibroblasts from Fibromuscular Dysplasia (FMD) patients as compared to carefully matched control subjects. While this remains among the objectives, the study has been expanded to undertake a fully powered cross-tissue systems genetics analysis of FMD, and now also the related arteriopathies spontaneous coronary artery dissection (SCAD) and cervical artery dissection (CvAD). The overall objective is to disclose the core biologic mechanisms of these disorders.

DETAILED DESCRIPTION:
Specific aims

* Specific aim 1: To establish a library of fibroblasts, DNA, plasma and serum from patients with FMD, SCAD and CvAD and unaffected healthy control subjects.
* Specific aim 2: To perform a fully powered cross-tissue systems analysis of the key regulatory gene networks and disease drivers underlying FMD, SCAD and CvAD.
* Specific aim 3: To cross-compare the molecular and genomic profiles of FMD, SCAD and CvAD to establish the degree of biologic similarity among these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and freely willing to participate. For patients < 18 years of age consent will be via parents.
* Fluency in either English or Spanish.
* Signed, informed consent
* For FMD, SCAD or CvAD subjects - a clinical diagnosis of FMD, SCAD or CvAD with fulfillment of standard diagnostic criteria.
* For healthy controls - no clinical features of FMD, SCAD or CvAD and absence of any major ongoing systemic disease including any condition requiring hospitalization, immune suppression, intravenous or injected medications or that result in functional impairment in the performance of activities of daily living. Healthy controls will be matched to enrolled FMD patients on the basis of gender and approximate age (within a 5 year window of another FMD subject).

Exclusion Criteria:

* Patients who have co-morbidities which reduces life expectancy to one year.
* Patients with any solid organ or hematological transplantation, or those in whom transplantation is considered.
* Active autoimmune disease.
* Illicit drug use.
* HIV positive.
* Prior malignancy.
* Any other form of vascular disease, including other arteriopathy coronary artery disease or peripheral vascular disease
* Family history of arteriopathy other than FMD, SCAD or CvAD (e.g. Ehlers-Danlos syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will enroll 200 FMD patients, 100 SCAD patients, and 100 CvAD patients at the Mount Sinai Hospital. 200 matched healthy controls will also be recruited to this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of regulatory gene networks | single time point at study enrollment
  The identification of regulatory gene networks, and their key drivers, underlying FMD, SCAD and CvAD

SECONDARY OUTCOMES:
Identification of molecular features | single time point at study enrollment
  To cross-compare the molecular features of FMD, SCAD and CvAD
Identification of genomic features | single time point at study enrollment
  To cross-compare the genomic features of FMD, SCAD and CvAD
RNA sequencing | single time point at study enrollment
  To define and compare the genomic (RNA sequencing) profile of fibroblasts from FMD, SCAD and CvAD subjects versus healthy control subjects
Circulating cytokine | single time point at study enrollment
  To define and compare the circulating cytokine profile of FMD versus healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kovacic, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jeffrey Olin, DO, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Olin JW, Di Narzo AF, d'Escamard V, Kadian-Dodov D, Cheng H, Georges A, King A, Thomas A, Barwari T, Michelis KC, Bouchareb R, Bander E, Anyanwu A, Stelzer P, Filsoufi F, Florman S, Civelek M, Debette S, Jeunemaitre X, Bjorkegren JLM, Mayr M, Bouatia-Naji N, Hao K, Kovacic JC. A plasma proteogenomic signature for fibromuscular dysplasia. Cardiovasc Res. 2020 Jan 1;116(1):63-77. doi: 10.1093/cvr/cvz219. PMID 31424497
- [Result] Kiando SR, Tucker NR, Castro-Vega LJ, Katz A, D'Escamard V, Treard C, Fraher D, Albuisson J, Kadian-Dodov D, Ye Z, Austin E, Yang ML, Hunker K, Barlassina C, Cusi D, Galan P, Empana JP, Jouven X, Gimenez-Roqueplo AP, Bruneval P, Hyun Kim ES, Olin JW, Gornik HL, Azizi M, Plouin PF, Ellinor PT, Kullo IJ, Milan DJ, Ganesh SK, Boutouyrie P, Kovacic JC, Jeunemaitre X, Bouatia-Naji N. PHACTR1 Is a Genetic Susceptibility Locus for Fibromuscular Dysplasia Supporting Its Complex Genetic Pattern of Inheritance. PLoS Genet. 2016 Oct 28;12(10):e1006367. doi: 10.1371/journal.pgen.1006367. eCollection 2016 Oct. PMID 27792790
- [Result] Adlam D, Olson TM, Combaret N, Kovacic JC, Iismaa SE, Al-Hussaini A, O'Byrne MM, Bouajila S, Georges A, Mishra K, Braund PS, d'Escamard V, Huang S, Margaritis M, Nelson CP, de Andrade M, Kadian-Dodov D, Welch CA, Mazurkiewicz S, Jeunemaitre X; DISCO Consortium; Wong CMY, Giannoulatou E, Sweeting M, Muller D, Wood A, McGrath-Cadell L, Fatkin D, Dunwoodie SL, Harvey R, Holloway C, Empana JP, Jouven X; CARDIoGRAMPlusC4D Study Group; Olin JW, Gulati R, Tweet MS, Hayes SN, Samani NJ, Graham RM, Motreff P, Bouatia-Naji N. Association of the PHACTR1/EDN1 Genetic Locus With Spontaneous Coronary Artery Dissection. J Am Coll Cardiol. 2019 Jan 8;73(1):58-66. doi: 10.1016/j.jacc.2018.09.085. PMID 30621952
- [Result] Georges A, Albuisson J, Berrandou T, Dupre D, Lorthioir A, D'Escamard V, Di Narzo AF, Kadian-Dodov D, Olin JW, Warchol-Celinska E, Prejbisz A, Januszewicz A, Bruneval P, Baranowska AA, Webb TR, Hamby SE, Samani NJ, Adlam D, Fendrikova-Mahlay N, Hazen S, Wang Y, Yang ML, Hunker K, Combaret N, Motreff P, Chedid A, Fiquet B, Plouin PF, Mousseaux E, Azarine A, Amar L, Azizi M, Gornik HL, Ganesh SK, Kovacic JC, Jeunemaitre X, Bouatia-Naji N. Rare loss-of-function mutations of PTGIR are enriched in fibromuscular dysplasia. Cardiovasc Res. 2021 Mar 21;117(4):1154-1165. doi: 10.1093/cvr/cvaa161. PMID 32531060